CLINICAL TRIAL: NCT02702895
Title: Assessment of ASPIRE and HOPE Adherence
Status: Completed | Type: Observational
Sponsor: Microbicide Trials Network (Network)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Other Study IDs: MTN-032; UM1AI068633 (NIH); UM1AI068615 (NIH); UM1AI106707 (NIH); Protocol ID#12058 (Other Grant/Funding Number: DAIDS)
Record Dates: First submitted 2015-08-31; First posted 2016-03-09 (Estimated); Last update posted 2022-10-13 (Actual); Status verified 2021-06

CONDITIONS: HIV Prevention

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Phase 1: Former ASPIRE participants
  Interventions: Behavioral: In-depth Interview (IDIs) or Focus Group Discussion (FGD)
- Phase 2 HOPE participants: Former HOPE participants
  Interventions: Behavioral: In-depth Interview (IDIs) or Focus Group Discussion (FGD)
- Phase 2 Male Partners: Male partners of HOPE participants
  Interventions: Behavioral: In-depth Interview (IDIs) or Focus Group Discussion (FGD)

INTERVENTIONS:
Behavioral: In-depth Interview (IDIs) or Focus Group Discussion (FGD)

SUMMARY:
MTN-032 is an exploratory sub-study of the ASPIRE and HOPE trials that will utilize qualitative In-Depth Interviews (IDIs) and Focus-Group Discussions (FGDs) to explore socio-contextual and trial specific issues which affected participants' adherence to the dapivirine vaginal ring (VR), as well as male partner attitudes towards and experiences with the dapivirine VR and their perspective of their female partner's attitudes and experiences.

DETAILED DESCRIPTION:
The MTN-032 trial is a two-phase exploratory sub-study of the ASPIRE and HOPE trials. A total of 187 former ASPIRE participants aged 19-48 years were enrolled in Phase 1 of this study. Up to 156 HOPE participants and up to 120 male partners of HOPE participants will be selected for participation in Phase 2 of this study. There were approximately 4-6 months allotted for recruitment and follow-up at each site for Phase 1, and 9-12 months allotted for recruitment and follow-up at each site for Phase 2..

MTN-032, an observational study, using interviews and focus group discussions, is primarily designed to identify factors that may have affected participant adherence to study product in ASPIRE and HOPE, including male partner attitudes. MTN-032 will also elicit perceptions about various participant engagement and adherence promotion interventions implemented in ASPIRE and may also explore the potential use of incentives to promote adherence to VR use.

MTN-032 will use study product adherence results from ASPIRE and HOPE, qualitative in-depth interviews (IDI) and focus group discussions (FGD) to explore study product adherence behaviors and strategies used to overcome adherence challenges. An in-depth understanding of the various socio-behavioral factors that contribute to product use adherence may assist in the interpretation of past and ongoing study results and inform implementation of future studies.

ELIGIBILITY:
Inclusion Criteria (Phase 1 - Former ASPIRE participants):

1. Participated in the ASPIRE protocol, randomized to active product and informed of their randomization assignment.
2. Able and willing to provide written informed consent in one of the study languages.
3. Able and willing to complete the required study procedures.
4. For participants who did not acquire an HIV infection while taking part in ASPIRE, evidence of study product dispensation at a minimum of three consecutive ASPIRE scheduled clinic visits. For participants who acquired an HIV infection while taking part in ASPIRE, evidence of study product dispensation in the month prior to the participant's acquisition of HIV infection.
5. For participants who did not acquire an HIV infection while taking part in ASPIRE, have a minimum of three ASPIRE PK data measurement points available. For participants who acquired HIV infection while taking part in ASPIRE, have a minimum of one ASPIRE PK data measurement available.

Inclusion Criteria (Phase 2 - HOPE participants):

1. Participated in the HOPE protocol.
2. Able and willing to provide written informed consent in one of the study languages.
3. Able and willing to complete the required study procedures.
4. For participants who did not acquire an HIV infection while taking part in HOPE, evidence of study product dispensation for a minimum of three consecutive months.
5. For participants who acquired an HIV infection while taking part in HOPE, evidence of study product dispensation in the month prior to the participant's acquisition of an HIV infection.

Inclusion Criteria (Phase 2 - Male partners of HOPE participants):

1. Identifies as a male sexual partner of a HOPE participant for whom the HOPE participant has given permission to contact.
2. Was a male sexual partner of a HOPE participant during her participation in HOPE (regardless of whether she used the ring or not).
3. Able and willing to provide written informed consent in one of the study languages.
4. Able and willing to complete the required study procedures.
5. Is above the age of 18 at the time of study participation.

Exclusion Criteria (Phase 1 and Phase 2):

1. Has any significant medical condition or other condition that, in the opinion of the Investigator of Record (IoR)/designee, would preclude informed consent, make study participation unsafe, complicate interpretation of study outcome data, or otherwise interfere with achieving the study objectives.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A sample of 187 former ASPIRE participants was selected to take part in Phase 1 of the study. A sample of up to 156 HOPE participants will be selected for participation in Phase 2. In addition, a sample of up to 120 male partners of HOPE participants who provided consent to have their male partners contacted will be selected for participation in Phase 2. Participants will all be adult women and their adult male partners from seven sites in three African countries: South Africa, Uganda and Malawi. It is anticipated that participants and their male partners will be representative of the overall ASPIRE and HOPE trials by enrolling participants from each of the participating ASPIRE and HOPE countries.
Sampling Method: Non-Probability Sample
Enrollment: 302 (Actual)
Dates: Start 2016-06-13 (Actual); Primary Completion 2018-12-19 (Actual); Study Completion 2019-12-19 (Actual)

PRIMARY OUTCOMES:
Factors affecting product use adherence | Phase 1: Four to six months during Q2/Q3 2016. Phase 2: Nine to twelve months during Q2 2018/Q2 2019.
  Socio-contextual and trial specific issues which affected participants' adherence to the dapivirine VR will be captured by IDI and/or FGD.
Male partner attitudes affecting product use adherence | Phase 2: Nine to twelve months during Q2 2018/Q2 2019.
  male partner attitudes towards and experiences with the dapivirine VR, and their perspective of their female partner's attitudes and experienceswill be captured by FGD and/or IDI.

SECONDARY OUTCOMES:
Perceptions of HIV risk | Phase 1: Four to six months during Q2/Q3 2016. Phase 2: Nine to twelve months during Q2 2018/Q2 2019.
  HIV risk and perceptions of HIV risk in general and specific to participants' and their male partners' motivation to participate in the ASPIRE and/or HOPE trial(s), to use study product (or not) during their participation in ASPIRE and/or HOPE, and male partner support (or lack thereof) of participants' product use in HOPE will be captured by IDI and/or FGD.
Product use patterns | Phase 1: Four to six months during Q2/Q3 2016. Phase 2: Nine to twelve months during Q2 2018/Q2 2019.
  Factors influencing product initiation and patterns of use during ASPIRE and/or HOPE will be captured by IDI and/or FGD.
Perceptions of various adherence support interventions | Phase 1: Four to six months during Q2/Q3 2016. Phase 2: Nine to twelve months during Q2 2018/Q2 2019.
  Participants' perceptions of various adherence support interventions and engagement activities implemented (or not implemented) during ASPIRE and/or HOPE will be captured by IDI and/or FGD.
Understanding of ASPIRE results and ring efficacy | Phase 1: Four to six months during Q2/Q3 2016. Phase 2: Nine to twelve months during Q2 2018/Q2 2019.
  Participants' and their male partners' understanding of the ASPIRE results and ring efficacy, and the impact of this understanding on participants' intention and/or ability to join HOPE and continue in follow-up, on their adherence to the dapivirine VR as part of an open label extension trial as compared to adherence in a Phase 3 safety and effectiveness trial, and male partner support (or lack thereof) of participants' trial participation and product use in HOPE will be captured by IDI and/or FGD.

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Montgomery, PhD, MHS, Study Chair — RTI International
Locations (7):
- Malawi Clinical Research Site, Lilongwe, Malawi
- South Africa (3):
  - Botha's Hill Clinical Research Site, Durban, KwaZulu-Natal
  - CAPRISA eThekwini Clinical Research Site, Durban, KwaZulu-Natal
  - Wits Reproductive Health and HIV Institute Clinical Research Site, Johannesburg
- Makerere University - Johns Hopkins University Research Collaboration Clinical Research Site, Kampala, Uganda
- Zimbabwe (2):
  - Spilhaus Clinical Research Site, Harare
  - Zengeza Clinical Research Site, Harare

REFERENCES:
- [Result] Montgomery ET, Stadler J, Naidoo S, Katz AWK, Laborde N, Garcia M, Reddy K, Mansoor LE, Etima J, Zimba C, Chitukuta M, Soto-Torres L. Reasons for nonadherence to the dapivirine vaginal ring: narrative explanations of objective drug-level results. AIDS. 2018 Jul 17;32(11):1517-1525. doi: 10.1097/QAD.0000000000001868. PMID 29957723
- [Result] Naidoo K, Mansoor LE, Katz AWK, Garcia M, Kemigisha D, Morar NS, Zimba CC, Chitukuta M, Reddy K, Soto-Torres L, Naidoo S, Montgomery ET. Qualitative Perceptions of Dapivirine VR Adherence and Drug Level Feedback Following an Open-Label Extension Trial. J Acquir Immune Defic Syndr. 2021 Apr 1;86(4):e90-e96. doi: 10.1097/QAI.0000000000002590. PMID 33278181
- [Result] Montgomery ET, Katz AWK, Duby Z, Mansoor LE, Morar NS, Naidoo K, Tsidya M, Chitukuta M, Guma V, Tenza S, Leslie J, Garcia M, Naidoo S. Men's Sexual Experiences with the Dapivirine Vaginal Ring in Malawi, South Africa, Uganda and Zimbabwe. AIDS Behav. 2021 Jun;25(6):1890-1900. doi: 10.1007/s10461-020-03119-2. Epub 2021 Jan 2. PMID 33389318